CLINICAL TRIAL: NCT05322551
Title: Molecular, Metabolomic and Nutritional Changes After Metabolic Surgery Among Obese Diabetic Patients and Biomarkers of Different Diabetes Status.
Brief Title: Molecular, Metabolomic and Nutritional Changes After Metabolic Surgery
Acronym: MoMen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Collaborators: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Fazliana Mansor, Research Officer, Ministry of Health, Malaysia
Other Study IDs: NMRR-20-2496-56353
Record Dates: First submitted 2021-12-07; First posted 2022-04-12 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Endocrine; Diabete Type 2; PreDiabetes
Keywords: Bariatric surgery; Metabolic surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected for serum/plasma during baseline and 6 & 12 month follow-up Adipose tissue (omentum, visceral) will be collected during surgery. Venous blood samples (20mL = 4 teaspoons) will be collected prior to surgery, 6 month and 1 year postoperatively. The plasma samples will be obtained by centrifugation at 800 g for 15 min, and the aliquots will be transferred to polypropylene tubes and stored at -80°C until they are assayed. Total RNA and miRNA will be isolated according to manufacturer instructions.
  The first morning urine samples (minimum 30mL) will be collected. Frozen tubes will be used and stored at -80 °C until processing for Nuclear Magnetic Resonance (NMR) analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese only: Definition of Obese:
  Body Mass Index ≥ 30kg/m^2 (WHO classification)
  Definition of Non Diabetes: Fasting Plasma Glucose (FPG) < FPG 100 mg/dL (5.6 mmol/L)
- Obese with prediabetes: Definition of Obese:
  Body Mass Index ≥ 30kg/m^2 (WHO classification)
  Definition of Prediabetes: FPG 100 mg/dL (5.6 mmol/L) to 125 mg/dL (6.9 mmol/L) (IFG) OR A1C 5.7-6.4% (39-47 mmol/mol)
- Obese with diabetes: Definition of Obese:
  Body Mass Index ≥ 30kg/m^2 (WHO classification)
  Definition of Diabetes: (American Diabetes Association, 2020) FPG ≥126 mg/dL (7.0 mmol/L). Fasting is defined as no caloric intake for at least 8 h.* OR A1C ≥6.5% (48 mmol/mol).

SUMMARY:
Obesity is a major risk factor for Type 2 Diabetes (T2D) and cardiovascular diseases, such as hypertension and dyslipidemia. Recently, weight loss surgery (i.e., metabolic or bariatric surgery) has been shown to result in very good long-term glycemic control in patients with T2D and obesity. However, knowledge and data on molecular levels and metabolomics are still limited. This study will fill in these gaps and provide potential biomarkers for T2D. Lifestyle and dietary practices (LDP) influence the clinical outcome and metabolites in T2D. Although the roles of LDP is critical in ensuring optimal clinical outcomes, data is still limited especially on relating the LDP and metabolomics in T2D.

DETAILED DESCRIPTION:
Study design

This is a prospective single centre study to explore molecular aspects and metabolomic changes among 102 obese individuals of different diabetes status, undergoing metabolic surgery, which is currently performed in Hospital Kuala Lumpur, Malaysia. Serial measurements of the selected markers will be made pre-operative (baseline), at 6 and 12 months follow up after surgery. Twenty (20) healthy individuals will be recruited as controls.

Study population

All subjects with obesity (Body Mass Index ≥ 30kg/m^2 [WHO classification])) and diagnosed with pre-diabetes, T2D and non-diabetic (healthy) who are undergoing metabolic surgery at Hospital Kuala Lumpur will be recruited.

All patients referred by endocrinologists who are eligible and fulfill the inclusion and exclusion criteria for metabolic surgery will be included in the study until the sample size is achieved. Routinely, all patients will need to pay a visit to the clinic at 1, 2, 4 weeks after surgery, then 3, 6, 9, 12, 18, 24 months and after that, a life-long annual visit. Therefore, visit 6- and 12-month will be utilized for study follow-ups.

Metabolic surgery

The two most standard metabolic surgical procedures performed at Hospital Kuala Lumpur are laparoscopic sleeve gastrectomy and laparoscopic Roux en Y gastric bypass (RYGB). All the procedures are performed laparoscopically using 5-ports technique.

ELIGIBILITY:
Inclusion Criteria:

Patients' Inclusion Criteria

* BMI > 30kg/m2
* Men and women
* Ages 18-65 years old
* Diabetes status (non diabetic, pre diabetes and diabetes)
* Patients who will undergo metabolic surgery

Healthy individuals' Inclusion Criteria

* BMI < 30kg/m2,
* Men and women
* Ages 18-65 years old
* No diabetes
* No pre diabetes
* No other co-morbidities (high total cholesterol, high triglycerides, high blood pressure)

Exclusion Criteria:

Patients' Exclusion Criteria

* BMI <30 kg/m2
* Use of medications that may affect body weight at screening or during a 3 month period prior
* Other medical conditions like Cushing's, acromegaly, Heart failure, Crohn's disease, etc
* Alcohol dependence

Healthy Individuals' Exclusion Criteria

* BMI > 30 kg/m2 (obese)
* BMI < 18.5 kg/m2 (underweight)
* Diabetes status (pre diabetes and diabetes)
* Use of medications that may affect body weight at screening or during a 3 month period prior
* Other co-morbidities (high total cholesterol, high triglycerides, high blood pressure, cancer)
* Other medical conditions like Cushing's, acromegaly, Heart failure, Crohn's disease, etc
* Alcohol dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects with obesity (Body Mass Index ≥ 30kg/m2 [WHO classification])) and diagnosed with pre-diabetes, T2D and non-diabetic (healthy) who are undergoing metabolic surgery at Hospital Kuala Lumpur will be recruited. Healthy individuals will be recruited as controls for reference range
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Body weight changes | 6 months
  Body weight changes
Body weight changes | 12 months
  Body weight changes
Body mass index (BMI) changes | 6 months
  Body mass index changes measured in kg/m^2 (weight in kilograms, height in meters)
Body mass index (BMI) changes | 12 months
  Body mass index changes measured in kg/m^2 (weight in kilograms, height in meters)
Body Fat Percentage changes | 6 months
  Body Fat Percentage changes measured in percentage
Body Fat Percentage changes | 12 months
  Body Fat Percentage changes measured in percentage
Fasting Blood Glucose changes | 6 months
  Fasting Blood Glucose changes measured in mmol/L
Fasting Blood Glucose changes | 12 months
  Fasting Blood Glucose changes measured in mmol/L
HbA1c changes | 6 months
  HbA1c changes measured in percentage
HbA1c changes | 12 months
  HbA1c changes measured in percentage
Changes of metabolites profile | 6 months
  Changes of serum diabetes-related metabolites using Nuclear Magnetic Resonance (NMR)
Changes of metabolites profile | 12 months
  Changes of serum diabetes-related metabolites using Nuclear Magnetic Resonance (NMR)
Changes in lipid related biochemical parameters | 6 months
  Changes in triglyceride, total cholesterol, LDL cholesterol, HDL cholesterol levels in mmol/L
Changes in lipid related biochemical parameters | 12 months
  Changes in triglyceride, total cholesterol, LDL cholesterol, HDL cholesterol levels in mmol/L

SECONDARY OUTCOMES:
Quality of Life changes | At baseline, month 6 and month 12
  Quality of Life score measured by Obesity and Weight-Loss Quality of Life (OWLQOL ) questionnaire
Dietary Intake changes | At baseline, month 6 and month 12
  Dietary intake changes measured by Food Frequency Questionnaire (FFQ)

CONTACTS AND LOCATIONS:
Overall Officials: Fazliana Mansor, PhD, Principal Investigator — Institute for Medical Research, Setia Alam, Malaysia
Locations (1):
- Institute for Medical Research, National Institutes of Health, Shah Alam, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided